CLINICAL TRIAL: NCT05924022
Title: Hyperbaric Oxygen Treatment (HBOT) During Methadone Tapering in Human Subjects With Opioid Use Disorder
Brief Title: Hyperbaric Oxygen Treatment (HBOT) During Methadone Tapering
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Washington State University (Other)
Responsible Party: Principal Investigator, Marian Wilson, Associate Professor, Washington State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 20000
Record Dates: First submitted 2023-06-16; First posted 2023-06-29 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into 1 of 2 trial arms that will receive: 1) a 2-day medically-supervised full-dose HBOT treatment, or 2) a 2-day sub-therapeutic dose HBOT condition as a placebo control. Both groups will be receiving standard of care for addiction withdrawal symptoms, as managed and provided by their clinic physician and neither the full or sub-therapeutic HBOT dose are expected to affect their ongoing treatment. Updated to 3 arms 11/23/24: Participants will be randomized into one of three trial arms: (active arm of n = 12 in HBOT 100% oxygen and 2.0 ATA, active arm of n = 12 in HBOT 100% oxygen and 1.3 ATA, and sham arm of n = 12 in HBOT 21% oxygen and 1.3 ATA). All groups will be receiving standard of care for addiction withdrawal symptoms, as managed and provided by their clinic physician and neither the full or sub-therapeutic HBOT dose are expected to affect their ongoing treatment.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Only the HBOT personnel will be aware of the treatment assignments; the rest of the research team and participants will be blinded to condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Full treatment (Experimental): Participants are administered 100% oxygen in the HBOT chamber at 2.0 ATA
  Interventions: Combination Product: Hyperbaric Oxygen Treatment Full
- Partial pressure treatment (Active Comparator): Participants are administered 100% oxygen in the HBOT chamber at 1.3 ATA
  Interventions: Combination Product: Hyperbaric Oxygen Treatment Partial Pressure
- Sham (Sham Comparator): Participants are administered 21% oxygen n the HBOT chamber at 1.3 ATA.
  Interventions: Combination Product: Hyperbaric Oxygen Treatment Sham

INTERVENTIONS:
Combination Product: Hyperbaric Oxygen Treatment Full — Participants in this active treatment arm of the protocol will receive Hyperbaric Oxygen Treatment (HBOT)100% oxygen and 2.0 ATA prior to and the day of medically supervised 5% methadone dose reductions while sitting in a wheelchair-accessible, multi-place sealed pressurized chamber for 90 minutes each session.
  Arms: Full treatment
Combination Product: Hyperbaric Oxygen Treatment Sham — Participants in the sham condition arm of the protocol will receive Hyperbaric Oxygen Treatment (HBOT) 21% oxygen and 1.3 ATA prior to and the day of medically supervised 5% methadone dose reductions while sitting in a wheelchair-accessible, multi-place sealed pressurized chamber for 90 minutes each session receiving less than a fully pressurized 100% oxygen dose.
  Arms: Sham
Combination Product: Hyperbaric Oxygen Treatment Partial Pressure — Participants in this partial treatment arm of the protocol will receive Hyperbaric Oxygen Treatment (HBOT)100% oxygen and 1.3 ATA prior to and the day of medically supervised 5% methadone dose reductions while sitting in a wheelchair-accessible, multi-place sealed pressurized chamber for 90 minutes each session.
  Arms: Partial pressure treatment

SUMMARY:
The aims of this study are to 1) explore the efficacy of hyperbaric oxygen therapy (HBOT) applied at two different pressures compared to sham treatment in relieving signs and symptoms (both physical and psychological) of opioid withdrawal in human subjects associated with methadone dose reductions; and 2): explore whether HBOT can increase the odds of successful methadone dose reduction in patients who are interested in tapering their opioid dose. The investigators aim to explore, through qualitative methods, individual's experiences with treatment for opioid use disorder (OUD).

DETAILED DESCRIPTION:
The investigators will conduct a prospective, randomized, sham treatment-controlled trial to examine the efficacy of HBOT for improving signs and symptoms of opioid withdrawal in methadone-maintained OUD patients as they undergo two planned methadone dose reductions spaced two weeks apart.

A participant sample size of 24 was chosen based on power analysis guided by the investigators' earlier study that indicate that clinically meaningful results can be found with a minimum of 8 per group related to variables of highest interest i.e., pain and withdrawal symptoms.

Additionally to this trial, participants will be asked to partake in a semi-structured interview in which they will be asked to discuss (1) Beginning Treatment, (2) Life in Recovery, and (3) HBOT & Further Treatment.

Edited 11/23/24: An additional study arm was added to better address the question about the level of HBOT needed for effects. The new participant sample size of 36 was chosen based on power analysis guided by our earlier study that indicate that clinically meaningful results can be found with a minimum of 8 per group related to variables of highest interest i.e., pain and withdrawal symptoms. Participants will be randomized into one of three trial arms: (active arm of n = 12 in HBOT 100% oxygen and 2.0 ATA, partial active arm of n = 12 in HBOT 100% oxygen and 1.3 ATA, and sham arm of n = 12 in HBOT 21% oxygen and 1.3 ATA). All groups will be receiving standard of care for addiction withdrawal symptoms, as managed and provided by their clinic physician and neither the full or sub-therapeutic HBOT dose are expected to affect their ongoing treatment.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in a supervised opioid treatment program at the Spokane Regional Health District
* Age greater than 18 years
* Ability to read, speak, and write English
* Ability to provide written informed consent.

Exclusion Criteria:

* Pregnancy
* Any other medical or psychiatric condition that the PI, Co-PI (physician of record) or the Spokane Hyperbaric Center medical director determine might compromise safe study participation in the HBOT clinic (including but not limited to active psychosis, history of frequent psychiatric hospitalizations, severe anxiety with claustrophobia, aggression)
* Upper respiratory infection
* Emphysema
* Air cysts in the lung
* History of thoracic or ear surgery
* Taking the medication Antabuse for alcohol addiction
* High fever.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Adjective Rating Scale of Withdrawal (ARSW) | Subjects will be assessed for withdrawal signs and symptoms at week 1 and compared with the end of week 4.
  Self-reported opioid withdrawal symptoms will be captured using an online survey and compared from week 1 to week 4 timepoint. Score is summed from 16 items with a possible range of 0 to 144.

SECONDARY OUTCOMES:
Change in Methadone dose | The investigators will capture clinical chart dose records at one month and three months from baseline to determine if change in methadone was sustained
  The study design is for two 5% methadone dose reductions spaced two weeks apart to examine whether treatment group is better able to sustain the reduction.

CONTACTS AND LOCATIONS:
Overall Officials: Layton Matt, MD, Principal Investigator — Washington State University
Locations (1):
- Spokane Regional Health District, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: No